CLINICAL TRIAL: NCT05480449
Title: Phase 1/2b Trial of Autologous Humanized CD19-Directed Chimeric Antigen Receptor T-Cells Manufactured Using the CliniMACS Prodigy Platform for the Treatment of Pediatric B Cell Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: Autologous HuCART19 T Cells Manufactured Using the CliniMACS Prodigy Platform for Pediatric B-ALL (huCART19 Prodigy)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stephan Grupp MD PhD (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor-Investigator, Stephan Grupp MD PhD, Chief, Cell Therapy and Transplant Section Director, Susan S. and Stephen P. Kelly Center for Cancer Immunotherapy Medical Director, Cell and Gene Therapy Lab, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-019978; 22CT011 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: B Cell Acute Lymphoblastic Leukemia (B-ALL); B Lineage Lymphoblastic Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Arm (Experimental): The phase 1 dose escalation portion of the trial will use a standard "3+3" design to establish the recommended phase 2 dose of huCART19 cells in patients with subjects with prior treatment with CD19-directed CAR T cells. Two dose escalations of huCART19 are planned for the dose escalation phase.
  Interventions: Biological: Autologous Humanized CD19-Directed Chimeric Antigen Receptor T-Cells (huCART19)
- Dose Expansion Arms (Experimental): If at least one dose level of the dose escalation phase is determined to be safe, the phase 2b dose expansion phase of the trial will be opened to enrollment. Subjects will receive the highest dose of huCART19 cells that were determined to be safe in the dose escalation part of the trial. 2 cohorts are planned:
  * Cohort A (relapsed/refractory, CAR T cell naïve)
  * Cohort B (prior treatment with CD19-directed CAR T cells)
  Interventions: Biological: Autologous Humanized CD19-Directed Chimeric Antigen Receptor T-Cells (huCART19)

INTERVENTIONS:
Biological: Autologous Humanized CD19-Directed Chimeric Antigen Receptor T-Cells (huCART19) — The investigational agent in this protocol is humanized CART19 cells (huCART19). Autologous T cells will be engineered to express an extracellular single chain antibody (scFv) with specificity for CD19. This will be expected to redirect specificity of the transduced T cells for cells that express CD19, a molecule that is restricted in expression on the surface of the malignant cells and on normal B cells.

SUMMARY:
This study will determine the safety and efficacy of moving to a second-generation manufacturing process using the CliniMACS Prodigy platform to manufacture huCART19 cells for patients with B cell Acute Lymphoblastic Leukemia (B-ALL).

DETAILED DESCRIPTION:
Chimeric Antigen Receptor T-Cells (CAR T) cell therapy has shifted the treatment landscape for pediatric and young adult patients with multiply relapsed and refractory B-ALL (B cell Acute Lymphoblastic Leukemia), however, the manufacturing process remains in its first generation: laborious, time-intensive, and not automated. The time and significant personnel resources in this process can result in patient safety issues - with patients growing sicker, with harder to control leukemias - in the waiting period between T cell collection and completed CAR T cell product manufacture. Use of the CliniMACS Prodigy platform, that allows for semi-automated clinical-scale processing of huCART19 cell products in a functionally closed, sterile system, rapidly, without many of the logistical burdens encountered in the first-generation manufacturing method, can help to surmount these issues. This study will determine the safety and efficacy of moving to a second-generation manufacturing process using the CliniMACS Prodigy platform to manufacture huCART19 cells.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Informed Consent
2. Subjects with documented CD19+ ALL or Lly:

   a. Cohort A: Subjects with relapsed or refractory ALL or Lly who have not previously received CAR T-cell Therapy: i. 2nd or greater relapse (marrow or extramedullary) OR ii. Any relapse after allogeneic HSCT and ≥4 months from HSCT at enrollment OR iii. Refractory disease defined as having not achieved an MRD-negative (by multiparameter flow cytometry) or CSF-negative CR after ≥2 chemotherapy regimens/cycles of frontline therapy, or 1 cycle of reinduction therapy for subjects in first relapse OR iv. Newly diagnosed NCI high-risk B-ALL with induction failure, defined as a M3 bone marrow (≥25%) blasts at the end of induction chemotherapy OR v. First bone marrow relapse of B-ALL at <36 months after initial diagnosis OR vi. First or greater CNS relapse of B-ALL vii. Ineligible for allogeneic HSCT because of at least one of the following:

1. Comorbid disease 2. Other contraindications to HSCT conditioning regimen 3. Lack of suitable donor 4. Prior HSCT 5. Declines HSCT as the therapeutic option after documented discussion, with expected outcomes, and the role of HSCT with a BMT physician not a part of the study team.

b. Cohort B: Subjects with poor response to prior B cell directed engineered cell therapy, defined as any one of the following: i. Partial response or no response to prior cell therapy ii. CD19+ relapse after prior cell therapy, defined as bone marrow blasts > 0.01% by multiparameter flow cytometry or evidence of extramedullary disease iii. Demonstrated early (≤6 months from infusion) B cell recovery suggesting loss of engineered cells

3. Subjects with prior or current history of CNS3 disease will be eligible if Central Nervous System (CNS) disease is responsive to therapy.

4. Documentation of CD19 tumor expression in bone marrow, peripheral blood, cerebrospinal fluid (CSF), or tumor tissue by flow cytometry. If the subject has received CD19-directed therapy, flow cytometry should be obtained after this therapy to demonstrate CD19 expression.

5. Age 0-29 years

6. Adequate organ function.

a. Serum creatinine based on age/gender b. Adequate liver function: i. ALT within 5x ULN in the absence of ALL infiltration of the liver ii. Bilirubin ≤3x the upper limit of normal iii. ALT and/or bilirubin results that exceed this range are acceptable if, in the opinion of the physician-investigator (or as confirmed by liver biopsy), the abnormalities are directly related to ALL infiltration of the liver.

c. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and < Grade 3 hypoxia; DLCO ≥ 40% (corrected for anemia if necessary) if PFTs are clinically appropriate as determined by the investigator.

d. Left Ventricular Shortening Fraction (LVSF) ≥28% or Ejection Fraction (LVEF) ≥45% confirmed by echocardiogram or another scan. In cases where quantitative assessment of LVSF/LVEF is not possible, a statement by the cardiologist that the ECHO shows qualitatively normal ventricular function will suffice.

7. Adequate performance status defined as Lanksy or Karnofsky performance score ≥50

8. Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria:

1. Active hepatitis B or active hepatitis C
2. HIV infection
3. Active acute or chronic graft-versus-host disease (GVHD) requiring systemic therapy.
4. Concurrent use of systemic steroids or immunosuppression at the time of cell infusion or cell collection, or a condition, in the treating physician's opinion, that is likely to require steroid therapy or immunosuppression during collection or after infusion. Steroids for disease treatment at times other than cell collection or at the time of infusion are permitted. Use of physiologic replacement hydrocortisone or inhaled steroids is permitted as well.
5. CNS disease that is progressive on therapy, or with CNS parenchymal lesions that might increase the risk of CNS toxicity.
6. Subjects who are pregnant or nursing.
7. Uncontrolled active infection.
8. History of seizure disorder that requires ongoing anti-epileptic therapy.
9. If the subject has received previous CAR T cell therapies, history of grade 3 or higher ICANS following administration of a CAR T cell product.

Ages: 0 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 89 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2027-09-20 (Estimated); Study Completion 2029-09-20 (Estimated)

PRIMARY OUTCOMES:
Safety of huCART19 Administration | 5 years
  The safety of the administering Humanized Cd19-Directed Chimeric Antigen Receptor T-Cells (huCART9) will be measured by the monitoring the frequency and severity of adverse events in patients with advanced or refractory CD19+ hematologic malignancies, including those previously treated with cell therapy.
Efficacy of huCART19 Administration | 5 years
  The efficacy of huCART9 will be measured by the evaluating the overall response rate in patients with advanced or refractory CD19+ hematologic malignancies, including those previously treated with cell therapy.

SECONDARY OUTCOMES:
Manufacturing Feasibility | 5 years
  Manufacturing feasibility will be measured by the percentage of manufactured products that do not meet release criteria for vector transduction efficiency, T cell product purity, viability, sterility, or due to tumor contamination.
Safety of huCART19 as measured by ≥ Grade 3 toxicity rate | 5 years
  Safety of huCART19 as measured by ≥ Grade 3 toxicity rate (toxicity that is possibly attributed to huCART19) that is unmanageable, unexpected, and unrelated to chemotherapy.
Anti-tumor response due to huCART19 cell infusions | 5 years
  For subjects with detectable disease, measure anti-tumor response due to huCART19 cell infusions, as defined by the presence of medullary (morphologic or Minimal Residual Disease (MRD-level disease) and/or extramedullary disease at 1-month post-infusion.
Remission Rate | 5 years
  Overall remission rate will be measured by the proportion of treated subjects who achieve complete morphologic remission at Day 28 post huCART19 infusion.
huCART19 cell persistence | 5 years
  huCART 19 cell persistence will be measured by PCR (or flow) analysis of whole blood to detect and quantify survival of huCART19 cells over time.
Event Free Survival | 5 years
  1-year Event-Free Survival (EFS) in subjects with relapsed/refractory B-ALL (Cohort A) and in subjects with poor response to prior B cell directed engineered cell therapy (Cohort B).
Relapse-Free Survival | 5 years
  1-year Relapse-Free Survival (RFS) in subjects with relapsed/refractory B-ALL (Cohort A) and in subjects with poor response to prior B cell directed engineered cell therapy (Cohort B).
Overall Survival | 5 years
  1-year Overall Survival (OS) in subjects with relapsed/refractory B-ALL (Cohort A) and in subjects with poor response to prior B cell directed engineered cell therapy (Cohort B).

CONTACTS AND LOCATIONS:
Overall Officials: Allison Barz Leahy, MD, Principal Investigator — Children's Hospital of Philadelphia; Stephan Grupp, MD,PhD, Study Director — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States